CLINICAL TRIAL: NCT01814982
Title: An Open-Label, Single and Repeat Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-17299425 in Patients With Traumatic Brain Injury
Brief Title: An Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics Study of JNJ-17299425 in Participants With Traumatic Brain Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: reprioritization of company activities
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012997; 2007-000280-17 (EudraCT Number); 17299425TRM2001
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; JNJ-17299425; Intracranial pressure; Intravascular bolus injection
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1: JNJ-17299425 (Experimental): JNJ-1729425 will be administered once as 1 milligram (10 milliliter of a 0.1 milligram/milliliter (mg/ml) solution) intravenous bolus injection over 2 minutes in central vein. In case of no toxicity or Intra cranial pressure response, dose will be increased to a maximum of 200 milligram (mg).
  Interventions: Drug: JNJ-17299425
- Part 2: JNJ-17299425 (Experimental): JNJ-1729425 will be repeated once at a dose (which is, determined by Investigator in Part 1) as intravenous bolus injection over 2 minutes in central vein.
  Interventions: Drug: JNJ-17299425

INTERVENTIONS:
Drug: JNJ-17299425 — JNJ-17299425 will be administered at a starting dose of 1 milligram (10 milliliter of a 0.1 mg/ml solution) as intravenous bolus injection over 2 minutes in central vein.

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics (explores what the body does to the drug) and pharmacodynamics (the study of the action or effects a drug has on the body) of JNJ-17299425 in participants with traumatic brain injury (acute and chronic injuries to the brain, including the cerebral hemispheres, cerebellum, and brain stem).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (conducted in more than one center), and exploratory study of single and repeat, escalating, intravenous (injection of a substance into a vein) doses of JNJ-17299425 in participants with traumatic brain injury. The study consists of 2 parts (Part 1 and Part 2), and each part will have 2 stages (Stage 1 and Stage 2). In Stage 1 of each part only standard care will be given, through sedation, analgesia and ventilation. If Intra cranial pressure (ICP) rises to greater than 20 millimeter of mercury (mmHG) after ventricular drainage, participants will enter Stage 2 of each part and will receive JNJ-17299425 (single dose in Part 1 and repeated dose in Part 2). During Part 1, safety and efficacy of JNJ-17299425 will be evaluated and during Part 2, safety, tolerability, pharmacokinetics and pharmacodynamics of repeated doses will be evaluated. Efficacy will primarily be evaluated by reduction in ICP. Blood samples will be collected for pharmacokinetic evaluation at pre and post administration of study treatment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with traumatic head injury and requiring intracranial pressure (ICP) monitoring
* Post menopausal females, (or when known not to have menstruated for at least 12 months), or previously documented sterilization
* Body Mass Index (BMI=weight per square height): 18 to 35 kilogram per square meter inclusive
* Legally acceptable representatives (relatives or guardians) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are allowing the participant to participate in the study
* To participate in the optional pharmacogenomic component of this study, legally acceptable representatives (relatives or guardians) must have signed the informed consent form for pharmacogenomic research indicating willingness to participate in the pharmacogenomic component of the study (where local regulations permit). Refusal to consent for this component does not exclude a participant from participation in the clinical study

Exclusion Criteria:

* Major injury (multi-trauma) or disease outside the central nervous system causing significant vital organ or blood counts dysfunction (for example, disseminated intravascular coagulation, serious hepatic or kidney failure, acute respiratory distress syndrome, etc)
* Participants who already received specific ICP lowering therapy, other than ventricular drainage, before being dosed with JNJ-17299425
* Rapid increase of ICP expected to result in death of the participant
* Relevant abnormal values for hematology, clinical chemistry or urinalysis at admission
* Any known significant history or family history of anemia, hemolytic or autoimmune disease or thrombocytopenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Percentage Reduction in Intracranial Pressure (ICP) | 30 minutes post administration of JNJ-17299425
  The ICP is defined as the pressure within the cranial cavity. It is influenced by brain mass, the circulatory system, cerebrospinal fluid dynamics, and skull rigidity. Percentage reduction in ICP and reduction in ICP below 20 millimeter of mercury (mmHG) and a reduction of at least 15 percent ICP will be evaluated. Percentage reduction in ICP means ICP value at Baseline minus ICP value post administration of JNJ-17299425, divided by 100.
Absolute Intracranial Pressure (ICP) Reduction | 30 minutes post administration of JNJ-17299425
  Absolute ICP reduction is defined as difference between pre dose ICP and lowest ICP value achieved where ICP is pressure within cranial cavity.
Duration To Achieve ICP Reduction | 30 minutes post administration of JNJ-17299425
  Duration to achieve ICP reduction will assess the time at which ICP value is less than 20mmHg, and the time to achieve 50 percent and below 50 percent of absolute ICP reduction, and time at which lowest ICP value is achieved. Percentage reduction in ICP means ICP value at Baseline minus ICP value post administration of JNJ-17299425, divided by 100 and absolute ICP reduction is defined as difference between pre dose ICP and lowest ICP value achieved where ICP is pressure within cranial cavity.

SECONDARY OUTCOMES:
JNJ-17299425 Plasma Concentration | Pre dose and 2, 5, 10, 30 minutes and 1, 2, 3, 4, 6, 9, 12, 24, 36, 48 and 72 hours post administration of JNJ-17299425
  Plasma concentration of JNJ-17299425 will be determined by collecting venous blood samples at the defined time points.
Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Post Dose (AUC [0-24]) | Pre dose and 2, 5, 10, 30 minutes and 1, 2, 3, 4, 6, 9, 12, 24, 36, 48 and 72 hours post administration of first dose of JNJ-17299425, and at pre dose and 0.5, 1, 2, 3 and 12 hours post administration of second dose of JNJ-17299425
  The AUC (0-24) is the area under the plasma concentration-time curve from 0 to 24 hours post dosing.
Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Last Quantifiable Concentration (AUC[0-t]) and AUC From Time 0 to Infinite time (AUC ([0-infinity]) | Pre dose and 2, 5, 10, 30 minutes and 1, 2, 3, 4, 6, 9, 12, 24, 36, 48 and 72 hours post administration of first dose of JNJ-17299425, and at pre dose and 0.5, 1, 2, 3 and 12 hours post administration of second dose of JNJ-17299425
  The AUC (0-infinity) calculated by trapezoidal summation (time t is the time of the last quantifiable concentration C[last]) and AUC (infinity) is the area under the plasma concentration-time curve from time 0 to infinite time, calculated as the sum of AUC(last) and C(last)/l(z), in which C(last) is the last observed quantifiable concentration.
Clearance | Pre dose and 2, 5, 10, 30 minutes and 1, 2, 3, 4, 6, 9, 12, 24, 36, 48 and 72 hours post administration of first dose of JNJ-17299425, and at pre dose and 0.5, 1, 2, 3 and 12 hours post administration of second dose of JNJ-17299425
  Clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Volume of Distribution (V[d]) | Pre dose and 2, 5, 10, 30 minutes and 1, 2, 3, 4, 6, 9, 12, 24, 36, 48 and 72 hours post administration of first dose of JNJ-17299425, and at pre dose and 0.5, 1, 2, 3 and 12 hours post administration of second dose of JNJ-17299425
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Elimination Rate Constant (Lambda[z]) | Pre dose and at 2, 5, 10, 30 minutes and at 1, 2, 3, 4, 6, 9, 12, 24, 36, 48 and 72 hours after first dose and at pre dose and post administration of second dose, at 0.5, 1, 2, 3 and 12 hours after second dose of JNJ-17299425
  Lambda(z) determined by linear regression of the terminal points of the log-linear plasma concentration-time curve
Terminal Half-Life (t[1/2]) | Pre dose and 2, 5, 10, 30 minutes and 1, 2, 3, 4, 6, 9, 12, 24, 36, 48 and 72 hours post administration of first dose of JNJ-17299425, and at pre dose and 0.5, 1, 2, 3 and 12 hours post administration of second dose of JNJ-17299425
  Terminal half-life (t[(1/2]) is defined as 0.693/Lambda(z).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (11):
- Belgium (10):
  - Aalst
  - Brussels
  - Edegem
  - Genk
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
  - Roeselare
  - Turnhout
- Marseille, France